CLINICAL TRIAL: NCT00302198
Title: Amyotrophic Lateral Sclerosis Web Based Patient Care Database
Brief Title: Amyotrophic Lateral Sclerosis Web Based Patient Care Database: ALSConnection.Org
Status: Completed | Type: Observational
Sponsor: Forbes Norris MDA/ALS Research Center (Other)
Collaborators: Muscular Dystrophy Association (Other)
Other Study IDs: 23.112
Record Dates: First submitted 2006-03-10; First posted 2006-03-14 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-02

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Behavioral: ALS Registry

SUMMARY:
The purpose is to collect data for ALS research. The data will be used to learn more about the origin of ALS and to improve quality of care for people with ALS. The information you provide in the ALS registry will be used to evaluate variations in patient care, adherence to standards of care and also to help foster ALS research.

DETAILED DESCRIPTION:
Any person who has been diagnosed with ALS by a physician can enroll into this registry.

The information you provide in the ALS registry will be used to evaluate variations in patient care, adherence to standards of care and also to help foster ALS research. An additional focus of this website will be to educate participating patients and visitors to this site about ongoing ALS research.

ELIGIBILITY:
Inclusion Criteria:

* There are no inclusion and exclusion criteria beyond the fact that a person needs to have ALS in order to enroll.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient diagnosed with ALS by a licensed physician.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2006-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Miller, MD, Principal Investigator — California Pacific Medical Center
Locations (1):
- Forbes Norris MDA/ALS Center, San Francisco, California, United States